CLINICAL TRIAL: NCT07065357
Title: Treating the Metabolic Syndrome With a Sodium-glucose Cotransporter-2 Inhibitor: a Randomised Controlled Trial
Brief Title: Treating the Metabolic Syndrome With a Sodium-glucose Cotransporter-2 Inhibitor
Acronym: TIME-SGLT2
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN Yap Hang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 23-316
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Syndrome
Keywords: sodium-glucose cotransporter-2 inhibitor; metabolic syndrome; randomized controlled trial
MeSH Terms: conditions — Metabolic Syndrome | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2 inhibitor (Experimental)
  Interventions: Drug: Empagliflozin (oral)
- Placebo (Placebo Comparator)
  Interventions: Other: Matching placebo

INTERVENTIONS:
Drug: Empagliflozin (oral) — Participants received Empagliflozin 10 mg orally once daily for six months.
  Arms: SGLT2 inhibitor
Other: Matching placebo — Participants received matching placebo orally once daily for six months.
  Arms: Placebo

SUMMARY:
The metabolic syndrome occurs in overweight or obese people who also have abnormal lipids, blood pressure and blood glucose. It precedes the development of diabetes and cardiovascular complications. Currently, there are no drugs licensed for the treatment of the metabolic syndrome. Empagliflozin is a sodium-glucose cotransporter-2 (SGLT2) inhibitor, originally developed for diabetes but has since been proven to be beneficial in patients with heart and kidney failure. By increasing glucose excretion in the urine, it reduces body weight, body fat and blood pressure. The investigators therefore hypothesize that it may be the ideal drug to reverse the metabolic syndrome. Search of clinical trials registries shows that there are no industry sponsored trials targeting patients with the metabolic syndrome. The investigators propose to conduct a randomised controlled trial to study the effects of empagliflozin on 160 people with the metabolic syndrome, who will be randomised to receive either empagliflozin or placebo. The primary hypothesis is that empagliflozin will reduce the metabolic syndrome risk score, while secondary outcome measures include circulating levels of adipokines (adiponectin, fibroblast growth factor 21, adipocyte fatty acid-binding protein and lipocalin-2), body weight, waist circumference, blood pressure, glucose and lipids. This drug has already been approved for use in diabetes and cardiovascular risk prevention. This study, if positive, would provide evidence for its use in the metabolic syndrome and the treatment for this syndrome for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 18 years and younger than 85 years
* Fulfils the criteria for the metabolic syndrome [1] (waist ≥90cm in men or ≥80cm in women plus at least two other components: triglycerides ≥1.7 mmol/L; HDL <1.03 in men and <1.29 in women; blood pressure ≥130 mmHg systolic or ≥85 mmHg diastolic or previously diagnosed hypertension; fasting plasma glucose ≥5.6 mmol/L)
* Willing to take part in the study and give informed consent

Exclusion Criteria:

* Taking medications for diabetes, including oral agents, insulin or glucagon-like peptide-1 agonists
* Fasting plasma glucose ≥7.0 mmol/L or HbA1c ≥6.5% before randomisation
* Diagnosis of type 1 diabetes
* Taking medications for hypertension, unless the blood pressure is well controlled with a stable regime
* Patient who cannot be randomised to placebo because of a strong indication for an SGLT2 inhibitor
* Contraindications to empagliflozin (GFR <60 ml/min/1.73m2)
* History of intolerance or adverse reactions to an SGLT2 medication
* Co-morbidities that make the subject unsuitable to be a study subject
* Mental illness that makes the subject unsuitable
* Cognitive dysfunction
* Pregnancy
* Thyroid disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The change in the continuous metabolic syndrome risk score | From enrolment to the final visit at 6 months

SECONDARY OUTCOMES:
Serum level of adiponectin, AFABP, FGF21, lipocalin-2 | From enrolment to the final visit at 6 months
Body weight | From enrolment to the final visit at 6 months
Waist circumference | From enrolment to the final visit at 6 months
Sagittal abdominal diameter | From enrolment to the final visit at 6 months
Serum triglycerides | From enrolment to the final visit at 6 months
Serum HDL | From enrolment to the final visit at 6 months
Fasting glucose | From enrolment to the final visit at 6 months
HbA1c | From enrolment to the final visit at 6 months
HOMA2-IR | From enrolment to the final visit at 6 months
HOMA2-B | From enrolment to the final visit at 6 months
Systolic and diastolic blood pressure | From enrolment to the final visit at 6 months
The number of abnormal components of the metabolic syndrome in the subject | From enrolment to the final visit at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yap-Hang CHAN, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data that underlie the results reported in this publication.
Supporting Information: Study Protocol
Time Frame: after the publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee established for this purpose.